CLINICAL TRIAL: NCT07358338
Title: Application of Device-based Training to Improve Postural Control in Older Adults With Chronic Cerebral Ischemia
Brief Title: Application of Device-based Training to Improve Postural Control in Older Adults With CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Litvina Lyubov Dmitrievna (Other)
Responsible Party: Sponsor-Investigator, Litvina Lyubov Dmitrievna, physiotherapist, MEDSI Clinical Hospital 1, ICU
Organization: MEDSI Clinical Hospital 1, ICU (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32
Record Dates: First submitted 2025-12-25; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cerebrovascular Disorders; Gait Disorders, Neurologic; Accidental Fall; Aged; Postural Balance
MeSH Terms: conditions — Cerebrovascular Disorders; Gait Disorders, Neurologic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- training on the "Huber" (LPG-Systems, France) (Experimental): A course of treatments on the Huber stabilization trainer (LPG-Systems, France); a course of therapeutic exercises consisting of general strengthening exercises, as well as exercises aimed at improving balance and coordination; a course of massage of the cervical and shoulder area using a relaxing technique; a course of magnetic therapy (as indicated).
  Interventions: Device: "Huber" (LPG-Systems, France)
- treadmill training on the "C-mill" (Physiomed Elektromedizin AG, Germany) (Experimental): A course of treatments using a C-mill biofeedback video reconstruction treadmill (Physiomed Elektromedizin AG, Germany); a course of therapeutic exercises consisting of general strengthening exercises, as well as exercises aimed at improving balance and coordination; a course of massage of the cervical and shoulder area using a relaxing technique; a course of magnetic therapy (as indicated).
  Interventions: Device: "C-mill" (Physiomed Elektromedizin AG, Germany)
- Control group (Active Comparator): A course of therapeutic exercises consisting of general strengthening exercises, as well as exercises aimed at improving balance and coordination; a course of massage of the cervical and shoulder area using a relaxing technique; a course of magnetic therapy (as indicated).
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: "Huber" (LPG-Systems, France) — Procedures on the Huber stabilization trainer (LPG-Systems, France) include a 5-minute warm-up, followed by an individual selection of 3 tasks from the "Balance and Posture" program and 2 tasks from the "Resistance" program from levels 1 to 5.
  Arms: training on the "Huber" (LPG-Systems, France)
Device: "C-mill" (Physiomed Elektromedizin AG, Germany) — The procedures on the C-mill biofeedback video reconstruction track (Physiomed Elektromedizin AG, Germany) include a warm-up (3 minutes of normal walking), followed by blocks of tasks of 2-4 minutes each: "Slalom", "Tandem", "Obstacles", "Random Marks", "Speed Change", and ending with a cool-down (3 minutes of normal walking).
  Arms: treadmill training on the "C-mill" (Physiomed Elektromedizin AG, Germany)
Other: Physical therapy — The therapeutic exercise program consists of complex coordination exercises in various starting positions, including with objects. Each session will include a 5-minute warm-up, including breathing exercises and active joint exercises, followed by a 15-minute main block of exercises, and concludes with a 3-4-minute cool-down with stretching exercises for the back and lower extremities.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to improve comprehensive rehabilitation programs for elderly patients with chronic cerebral ischemia by incorporating training methods with biofeedback for postural control training.

The main objectives of the study are as follows:

To evaluate the effectiveness of incorporating stabilometric training with biofeedback using the Huber system (LPG Systems, France) and treadmill-based biofeedback training using the C-Mill system (Physiomed Elektromedizin AG, Germany) into comprehensive rehabilitation programs, with respect to postural and cognitive functions in elderly patients with chronic cerebral ischemia.

To conduct a comparative analysis of the effectiveness of training programs performed using the Huber (LPG Systems, France) and C-Mill (Physiomed Elektromedizin AG, Germany) biofeedback systems, based on outcomes related to gait pattern recovery, postural parameters, and cognitive performance.

The investigators will compare training sessions using the Huber and C-Mill biofeedback systems with a control group (patients receiving conventional therapeutic exercise) in order to determine whether these devices are effective in improving postural control and reducing the risk of falls in patients with chronic cerebral ischemia.

Participants are required to:

Complete a course consisting of 8 procedures, performed once daily. Report any adverse events occurring during or after the procedures, should they arise.

DETAILED DESCRIPTION:
This randomized controlled clinical study is designed to evaluate the effectiveness of biofeedback-based training methods incorporated into comprehensive rehabilitation programs for elderly patients with chronic cerebral ischemia.

The study population consists of patients aged 65 years and older with a confirmed diagnosis of chronic cerebral ischemia (ICD-10: I67.8) of atherosclerotic, hypertensive, or mixed etiology, presenting with clinical stage I or II disease and neuroimaging-confirmed structural brain changes. Participants will be randomized into three parallel groups with stratification to ensure comparability by age and severity of cognitive impairment.

Two intervention groups will receive standard inpatient rehabilitation combined with device-based training using biofeedback technologies. The first intervention group will undergo stabilometric training using the Huber system (LPG Systems, France), aimed at improving static and reactive components of postural control. The second intervention group will receive treadmill-based gait and balance training using the C-Mill system with visual biofeedback (Physiomed Elektromedizin AG, Germany), targeting dynamic balance, gait pattern restoration, and fall risk reduction. The control group will receive standard rehabilitation without device-based biofeedback training.

All participants will complete a comprehensive inpatient rehabilitation program lasting 10 days. Each program includes therapeutic exercise focused on general strengthening, balance, and coordination, as well as classical relaxing massage of the cervical-collar region and magnetotherapy when clinically indicated. Participants in the intervention groups will additionally complete 8 device-based training sessions. To ensure comparability across groups, the duration of active training time per session will be standardized and will range from 23 to 24 minutes.

Clinical and instrumental assessments will be conducted before and after the rehabilitation course to evaluate changes in postural stability, gait, mobility, cognitive function, fall risk, and quality of life. Fall risk will be assessed using the Morse Fall Scale, mobility using the Timed Up and Go Test, and cognitive function using the Montreal Cognitive Assessment. Instrumental evaluation of gait and balance will be performed using the C-Mill diagnostic C-Gait program, while postural and pedometric parameters will be assessed using the diagnostic module of the Huber system. Quality of life and psychological well-being will be evaluated using the EQ-5D-3L questionnaire.

The study hypothesizes that rehabilitation programs incorporating biofeedback-based device training will lead to more pronounced improvements in postural control, gait parameters, cognitive function, and fall risk reduction compared to conventional therapeutic exercise alone. It is expected that treadmill-based training using the C-Mill system will demonstrate a greater effect on dynamic balance and gait-related outcomes, whereas stabilometric training using the Huber system will primarily enhance static and reactive balance components. Improvements in quality of life are anticipated to be more pronounced in the biofeedback intervention groups.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly people aged 65 years and older, with a diagnosis of "Chronic cerebral ischemia" (according to the ICD-10 classification - I67.8 Other specified cerebral vascular lesions), atherosclerotic/hypertensive/mixed genesis (E.I. Gusev et al. 2022), clinical stage 1 or 2 according to the guidelines of the Research Institute of Neurology of the Russian Academy of Medical Sciences (2001) with neuroimaging-confirmed structural damage to the brain (stage 1 according to O.S. Levin (2006)
2. Signed voluntary consent to participate in the study.

Exclusion Criteria:

1. Age under 65, age over 98
2. Chronic diseases in the decompensation stage
3. Severe cognitive impairment
4. History of acute cerebrovascular accident
5. Presence of hemodynamically significant stenosis of the main cerebral arteries
6. Uncontrolled arterial hypertension
7. Neurodegenerative diseases
8. Dysmetabolic encephalopathy
9. History of traumatic brain injury
10. Condition after endoprosthetics of large joints
11. Severe sarcopenia
12. Oncological diseases in the progression stage
13. Lack of informed consent of the patient for the conduct of the study and access to information.

Ages: 65 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
The risk of falls was reduced more in groups using biofeedback equipment | 10 days
  Fall risk assessment using the Morse fall scale before and after the rehabilitation course (min 0, max 125, higher values on the scale indicate a worse outcome)
The risk of falls was reduced more in groups using biofeedback equipment | 10 days
  Fall risk assessment using the Get-Up-and-Go test before and after the rehabilitation course (Taking more than 14 seconds to complete the test indicates a high risk of falls)
The risk of falls was reduced more in groups using biofeedback equipment | 10 days
  Fall risk assessment using the gait speed before and after the rehabilitation course (a walking speed of more than 1 km/h indicates a high risk of falls)
Static balance will improve more in the group training on the "Huber", and dynamic balance in the group training on the treadmill "Cmill" | 10 days
  Evaluation based on the following stabilometric indicators: length and area of the statokinesiogram, average speed of oscillations of the body's center of pressure, indicators of the static and dynamic balance tests TUG, Romberg test with open and closed eyes, indicators of the dynamic walking stereotype (walking speed, step length, step variability)

SECONDARY OUTCOMES:
Improving cognitive functions | 10 days
  Montreal Cognitive Assessment (MoCA) (min 0 max 30 points, a higher score means a better result)
Improving the quality of life | 10 days
  EQ-5D-3L questionnaire (EuroQol five-dimension three-level questionnaire).The first part of the scale has a system of indices that form a code that does not calculate to a single score. The second part of the scale EQ VAS (scale from 0-100), has a range from 0 to 100, where 100 is the best state.

CONTACTS AND LOCATIONS:
Locations (1):
- MEDSI Clinic, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://panor.ru/articles/apparatnye-metodiki-trenirovki-dinamicheskikh-stereotipov-khodby-u-patsientov-starshikh-vozrastnykh-grupp/90324.html#
- See also: Related Info — http://cyberleninka.ru/article/n/vliyanie-stabilometricheskoy-platformy-na-snizhenie-riska-padeniy-u-pozhilyh-patsientov-s-hronicheskoy-ishemiey-golovnogo-mozga
- See also: Related Info — http://www.mediasphera.ru/issues/vosstanovitelnye-biotekhnologii-profilakticheskaya-tsifrovaya-i-prediktivnaya-meditsina/2024/2/13034252X2024021042